CLINICAL TRIAL: NCT03952377
Title: A Double-Blind, Randomized, Placebo-Controlled, Parallel-Group Phase I/II, First-in-Human Study to Assess the Safety and Efficacy of Two Doses of SX600 Administered by Lumbosacral Transforaminal Epidural Injection in Patients With Radicular Pain Secondary to Lumbar Intervertebral Disc Herniation
Brief Title: Safety and Efficacy of SX600 Administered by Lumbosacral Transforaminal Epidural Injection for Radicular Pain
Acronym: SALIENT
Status: Terminated | Phase: Phase 1 / Phase 2 | Type: Interventional
Why Stopped: Due to the impact of COVID-19 and associated enrollment difficulties, the study was terminated with a total sample size of 56 randomized patients
Sponsor: SpineThera Australia PTY LTD (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: CLIN-0012-STA19-01
Record Dates: First submitted 2019-05-13; First posted 2019-05-16 (Actual); Results first posted 2024-01-10 (Actual); Last update posted 2024-01-10 (Actual); Status verified 2023-12

CONDITIONS: Lumbar Radiculopathy
Keywords: Sciatica; Low Back Pain; Lumbosacral Radiculopathy; Leg Pain
MeSH Terms: conditions — Radiculopathy; Sciatica; Low Back Pain

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Masking Description: Double-Blind
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (3):
- 0.9% Sodium Chloride for Injection (Placebo Comparator)
  Interventions: Drug: Placebo
- 12.5 mg SX600 (Experimental): Low Dose
  Interventions: Drug: SX600
- 25.0 mg SX600 (Experimental): High Dose
  Interventions: Drug: SX600

INTERVENTIONS:
Drug: SX600 — Transforaminal Epidural Injection
  Arms: 12.5 mg SX600; 25.0 mg SX600
Drug: Placebo — Transforaminal Epidural Injection
  Arms: 0.9% Sodium Chloride for Injection

SUMMARY:
This is a Phase I/II, double-blind, parallel-group, randomized, placebo-controlled multi-centre trial in 180 patients randomized 1:1:1 to receive the IMP (Dexamethasone acetate microspheres for extended-release injectable micro-suspension, SX600 at 12.5 mg or 25.0 mg) or Placebo (0.9% Sodium Chloride for Injection, BP) via transforaminal epidural injection to the lumbosacral epidural space.

ELIGIBILITY:
Main Inclusion Criteria:

* Adult aged 18 to 65 years, capable of providing informed consent, capable of complying with the outcome instruments, and meeting the attendance requirements for review as defined in the study
* Presenting with a history of radicular pain of duration of 4 weeks to 6 months, having failed conservative therapy.
* Mean Worst Daily Leg Pain score of ≥5.0 and ≤9.0
* Women of child-bearing potential must use a medically accepted method of contraception for the duration of the study plus 30 days and register a negative pregnancy test prior to dosing

Main Exclusion Criteria:

* Documented history of allergy or intolerance to components of the Investigational Medicinal Product, relevant radiologic contrast media, or local anaesthetics
* Is pregnant or lactating
* Has been taking corticosteroid medications routinely in the past 6 months or has received an epidural corticosteroid injection within 12 weeks of screening
* Has a BMI greater than 40 kg/m2
* Has radiological evidence of clinically significant foraminal stenosis at L4-L5 or L5-S1 or of clinically significant spinal stenosis, or spondylolisthesis (Grade 2 or higher). (Note, asymptomatic foraminal stenosis at other spinal levels is not excluded).
* Has Diabetes Mellitus (Type 1 or Type 2)- prior confirmed HbA1c or OGTT
* Has a history of significant leg pain unrelated to disc herniation that would significantly compromise assessment of back or leg radicular pain
* Has had lumbar back surgery
* Has received an implantable device for pain management

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 56 (Actual)
Dates: Start 2019-11-04 (Actual); Primary Completion 2022-02-21 (Actual); Study Completion 2022-06-21 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Willem Volschenk, Principal Investigator — Genesis Research Services
Locations (10):
- Australia (10):
  - Research Site 03, Adelaide
  - Research Site 12, Adelaide
  - Research Site 10, Blacktown
  - Research Site 06, Frankston
  - Research Site 05, Newcastle
  - Research Site 02, Sydney
  - Research Site 04, Sydney
  - Research Site 09, Sydney
  - Research Site 11, Sydney
  - Research Site 08, Townsville

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | 0.9% Sodium Chloride for Injection | 12.5 mg SX600 | 25.0 mg SX600
Started | 18 | 21 | 17
Completed | 16 | 19 | 16
Not Completed | 2 | 2 | 1

BASELINE CHARACTERISTICS:
Population: ITT Population
Groups:
- Total: Total of all reporting groups
Arm/Group | 0.9% Sodium Chloride for Injection | 12.5 mg SX600 | 25.0 mg SX600 | Total
Number analyzed (Participants) | 18 | 21 | 17 | 56
Age, Continuous [Mean (Standard Deviation); unit: years] | 45.1 (6.77) | 47.7 (7.25) | 52.0 (4.86) | 48.1 (6.93)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 7 | 5 | 7 | 19
  Male | 11 | 16 | 10 | 37
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0
  Asian | 2 | 3 | 0 | 5
  Native Hawaiian or Other Pacific Islander | 1 | 0 | 0 | 1
  Black or African American | 0 | 0 | 0 | 0
  White | 13 | 17 | 14 | 44
  More than one race | 0 | 0 | 0 | 0
  Unknown or Not Reported | 2 | 1 | 3 | 6
Region of Enrollment [Number; unit: participants]
  Australia | 18 | 21 | 17 | 56

OUTCOME MEASURES:

1. Primary Outcome: The Proportion of Subjects With a 50% or Greater Improvement in Mean Worst Daily Leg Pain (Responders).
Time Frame: Baseline to 60 days
Population: mITT population, denominator (# of participants analyzed) is number of non-missing values at 60 days
Measure: Count of Participants; unit: Participants
Arm/Group | 0.9% Sodium Chloride for Injection | 12.5 mg SX600 | 25.0 mg SX600
Number analyzed (Participants) | 16 | 19 | 14
Participants | 2 | 10 | 10

2. Secondary Outcome: The Proportion of Subjects Who Are Responders (Defined as Having a 50% or Greater Improvement in Mean Worst Daily Leg Pain)
Time Frame: Baseline to 14, 30, 60, 90, 120, 150, and 180 days
Population: Denominator for % is the number of non-missing values for each treatment group at the visit of interest for the mITT population
Measure: Number; unit: percentage of participants
Arm/Group | 0.9% Sodium Chloride for Injection | 12.5 mg SX600 | 25.0 mg SX600
Number analyzed (Participants) | 18 | 21 | 16
percentage of participants
  Baseline to 14 days: number analyzed (Participants) | 18 | 19 | 16
  Baseline to 14 days | 22.2 | 42.1 | 43.8
  Baseline to 30 days: number analyzed (Participants) | 17 | 18 | 15
  Baseline to 30 days | 17.6 | 38.9 | 66.7
  Baseline to 90 days: number analyzed (Participants) | 16 | 19 | 15
  Baseline to 90 days | 43.8 | 52.6 | 66.7
  Baseline to 120 days: number analyzed (Participants) | 15 | 15 | 14
  Baseline to 120 days | 46.7 | 46.7 | 64.3
  Baseline to 150 days: number analyzed (Participants) | 12 | 15 | 14
  Baseline to 150 days | 41.7 | 46.7 | 71.4
  Baseline to 180 days: number analyzed (Participants) | 13 | 15 | 13
  Baseline to 180 days | 38.5 | 46.7 | 69.2

3. Secondary Outcome: Change in Functional Outcomes as Measured by Patient's Global Impression of Change
Description: Very much improved, or much improved from baseline
Time Frame: Baseline, 14, 30, 60, 90, 120, 150, and 180 days
Population: % based on number of non-missing values at the time of visit in mITT population
Measure: Number; unit: percentage of participants
Arm/Group | 0.9% Sodium Chloride for Injection | 12.5 mg SX600 | 25.0 mg SX600
Number analyzed (Participants) | 18 | 21 | 16
percentage of participants
  Baseline to 14 days: number analyzed (Participants) | 18 | 19 | 16
  Baseline to 14 days | 16.7 | 36.8 | 56.3
  Baseline to 30 days: number analyzed (Participants) | 17 | 20 | 15
  Baseline to 30 days | 23.5 | 45 | 53.3
  Baseline to 60 days: number analyzed (Participants) | 17 | 20 | 15
  Baseline to 60 days | 23.2 | 45 | 60
  Baseline to 90 days: number analyzed (Participants) | 16 | 18 | 15
  Baseline to 90 days | 50 | 38.9 | 60
  Baseline to 120 days: number analyzed (Participants) | 13 | 15 | 14
  Baseline to 120 days | 46.2 | 46.7 | 57.1
  Baseline to 150 days: number analyzed (Participants) | 12 | 15 | 14
  Baseline to 150 days | 58.3 | 46.7 | 57.1
  Baseline to 180 days: number analyzed (Participants) | 12 | 16 | 14
  Baseline to 180 days | 66.6 | 50.1 | 71.5

4. Secondary Outcome: Change in Functional Outcomes as Measured by the Oswestry Disability Index
Description: 0 - 20%: Minimal disability 21% - 40%: Moderate disability 41% - 60%: Severe disability 61% - 80%: Crippling back pain 81% - 100%: Bed-bound or exaggerating their symptoms
Time Frame: Baseline, 14, 30, 60, 90, 120, 150, and 180 days
Population: % based on number of non-missing values at the time of the visit for the mITT population
Measure: Mean (Standard Deviation); unit: score on scale of 0% to 100%
Arm/Group | 0.9% Sodium Chloride for Injection | 12.5 mg SX600 | 25.0 mg SX600
Number analyzed (Participants) | 18 | 21 | 16
score on scale of 0% to 100%
  Baseline: number analyzed (Participants) | 17 | 21 | 16
  Baseline | 27.99 (9.525) | 35.21 (12.844) | 32.83 (16.113)
  14 days: number analyzed (Participants) | 18 | 19 | 16
  14 days | 22.97 (12.730) | 21.04 (14.463) | 19.72 (19.506)
  30 days: number analyzed (Participants) | 17 | 20 | 15
  30 days | 19.22 (10.341) | 21.12 (16.464) | 16.89 (19.427)
  60 days: number analyzed (Participants) | 17 | 20 | 15
  60 days | 17.64 (11.306) | 16.50 (13.839) | 15.31 (19.237)
  90 days: number analyzed (Participants) | 16 | 18 | 15
  90 days | 17.06 (12.841) | 14.67 (10.847) | 16.95 (22.502)
  120 days: number analyzed (Participants) | 13 | 15 | 14
  120 days | 12.8 (8.193) | 16.53 (12.794) | 19.59 (24.574)
  150 days: number analyzed (Participants) | 12 | 15 | 14
  150 days | 11.89 (6.578) | 14.13 (11.426) | 12.74 (11.994)
  180 days: number analyzed (Participants) | 12 | 16 | 14
  180 days | 12.23 (7.208) | 15 (13.779) | 9.74 (8.781)

5. Secondary Outcome: Change From Baseline in Short Form 36 Questionnaire (SF-36)
Description: SF-36 is a self-administered, generic health status questionnaire consisting of 36 questions that measure 8 health concepts: physical functioning, bodily pain, role limitations due to physical health problems, role limitations due to personal or emotional problems, emotional well-being, social functioning, energy/fatigue, and general health perceptions. Each health concept has a range of possible total scores from 0 to 100. A high score defines a more favorable health state. The mean overall total score will be reported.
Time Frame: Baseline, 14, 30, 60, 90, 120, 150, and 180 days
Population: mITT population
Measure: Mean (Full Range); unit: score on a scale
Arm/Group | 0.9% Sodium Chloride for Injection | 12.5 mg SX600 | 25.0 mg SX600
Number analyzed (Participants) | 18 | 21 | 16
score on a scale
  Baseline | 61.03 [0 to 100] | 51.04 [0 to 100] | 48.40 [0 to 100]
  14 days: number analyzed (Participants) | 18 | 19 | 16
  14 days | 60.85 [0 to 100] | 63.73 [0 to 100] | 61.89 [0 to 100]
  30 days: number analyzed (Participants) | 17 | 20 | 15
  30 days | 64.02 [0 to 100] | 63.28 [0 to 100] | 67.93 [0 to 100]
  60 days: number analyzed (Participants) | 17 | 20 | 15
  60 days | 66.17 [0 to 100] | 73.26 [0 to 100] | 69.29 [0 to 100]
  90 days: number analyzed (Participants) | 16 | 18 | 15
  90 days | 69.07 [0 to 100] | 73.22 [0 to 100] | 68.8 [0 to 100]
  120 days: number analyzed (Participants) | 13 | 15 | 14
  120 days | 77.32 [0 to 100] | 69.49 [0 to 100] | 68 [0 to 100]
  150 days: number analyzed (Participants) | 12 | 15 | 14
  150 days | 73.92 [0 to 100] | 76 [0 to 100] | 72.44 [0 to 100]
  180 days: number analyzed (Participants) | 12 | 16 | 14
  180 days | 77.83 [0 to 100] | 72.57 [0 to 100] | 77.29 [0 to 100]

6. Secondary Outcome: The Proportion of Subjects Who Are Responders (Defined as Having a 30% or Greater Improvement in Mean Worst Daily Leg Pain)
Time Frame: Baseline to 14, 30, 60, 90, 120, 150, and 180 days
Population: mITT population
Measure: Number; unit: percentage of participants
Arm/Group | 0.9% Sodium Chloride for Injection | 12.5 mg SX600 | 25.0 mg SX600
Number analyzed (Participants) | 18 | 21 | 16
percentage of participants
  14 days: number analyzed (Participants) | 18 | 19 | 16
  14 days | 27.8 | 52.6 | 68.8
  30 days: number analyzed (Participants) | 17 | 18 | 15
  30 days | 29.4 | 61.1 | 80
  60 days: number analyzed (Participants) | 16 | 19 | 14
  60 days | 50 | 73.7 | 78.6
  90 days: number analyzed (Participants) | 16 | 20 | 15
  90 days | 50 | 60 | 66.7
  120 days: number analyzed (Participants) | 15 | 16 | 14
  120 days | 53.3 | 50 | 71.4
  150 days: number analyzed (Participants) | 13 | 16 | 14
  150 days | 46.2 | 62.5 | 71.4
  180 days: number analyzed (Participants) | 15 | 16 | 13
  180 days | 46.7 | 50 | 76.9

7. Secondary Outcome: Proportion of Subjects Who Required Rescue Medication, as Reported in Patient Diary
Time Frame: Baseline through 180 days
Population: ITT population
Measure: Count of Participants; unit: Participants
Arm/Group | 0.9% Sodium Chloride for Injection | 12.5 mg SX600 | 25.0 mg SX600
Number analyzed (Participants) | 18 | 21 | 17
Participants | 7 | 3 | 3

8. Secondary Outcome: Time to Loss of Response in the Subset of Patients Who Are Responders at Day 14 (50% or Greater Improvement in Mean Worst Daily Leg Pain)
Time Frame: Day 14 through 180 days
Population: Time to loss of response was analyzed in the subset of patients who had a 50% or greater improvement in mean WDLP score (i.e., 50% Responders) at Day 14 compared to Baseline.
Measure: Mean (Standard Error); unit: days
Arm/Group | 0.9% Sodium Chloride for Injection | 12.5 mg SX600 | 25.0 mg SX600
Number analyzed (Participants) | 4 | 8 | 7
days | 40.8 (7.54) | 40.8 (6.19) | 103.3 (2.24)

9. Other Pre Specified Outcome: Proportion of Subjects Who Reduce Utilization of Supportive Health Services From Baseline, as Reported in Patient Diary
Time Frame: From baseline through 180 days
Population: This endpoint was not included in the final SAP, thus this analysis was not conducted.
Arm/Group | 0.9% Sodium Chloride for Injection | 12.5 mg SX600 | 25.0 mg SX600
Number analyzed (Participants) | 0 | 0 | 0

ADVERSE EVENTS:
Time Frame: 180 days
Description: 1 of the 17 subjects in the 25 mg SX600 group did not receive the study drug due to the inability to complete the TF-EI procedure due to unsure transitional anatomy, thus was not included in the safety population. Participants at risk in this group is thus, 16 (not 17 as listed in participant flow).
Arm/Group | 0.9% Sodium Chloride for Injection | 12.5 mg SX600 | 25.0 mg SX600
All-Cause Mortality (participants affected / at risk) | 0/18 | 0/21 | 0/16
Serious Adverse Events (participants affected / at risk) | 3/18 | 0/21 | 1/16
Other Adverse Events (participants affected / at risk) | 15/18 | 16/21 | 14/16
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | 0.9% Sodium Chloride for Injection (N=18) | 12.5 mg SX600 (N=21) | 25.0 mg SX600 (N=16)
Small Intestinal Obstruction (Gastrointestinal disorders) | 1 | 0 | 0
Back Pain (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0
Radiculopathy (Nervous system disorders) | 1 | 0 | 0
Renal Colic (Renal and urinary disorders) | 0 | 0 | 1 — Based on Sponsor review of this case, this SAE may be more consistent with increased low back and radicular leg pain
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | 0.9% Sodium Chloride for Injection (N=18) | 12.5 mg SX600 (N=21) | 25.0 mg SX600 (N=16)
Alanine aminotransferase increased (Investigations) | 0 | 4 | 2
Blood cholesterol increased (Investigations) | 2 | 2 | 2
Blood creatine phosphokinase increased (Investigations) | 2 | 1 | 3
Blood lactate dehydrogenase increased (Investigations) | 2 | 1 | 2
Low density lipoprotein increased (Investigations) | 2 | 2 | 1
Aspartate aminotransferase increased (Investigations) | 0 | 0 | 2
Bilirubin conjugated increased (Investigations) | 2 | 0 | 0
Blood bilirubin increased (Investigations) | 2 | 0 | 0
Blood uric acid increased (Investigations) | 1 | 0 | 1
Gamma-glutamyltransferase increased (Investigations) | 0 | 2 | 0
White blood cell count increased (Investigations) | 0 | 1 | 1
Blood fibrinogen increased (Investigations) | 0 | 0 | 1
Blood glucose decreased (Investigations) | 1 | 0 | 0
Blood pressure increased (Investigations) | 0 | 0 | 1
Blood triglycerides increased (Investigations) | 1 | 0 | 0
Blood urine present (Investigations) | 0 | 0 | 1
Eosinophil count increased (Investigations) | 1 | 0 | 0
Glomerular filtration rate decreased (Investigations) | 1 | 0 | 0
Hepatic enzyme increased (Investigations) | 0 | 0 | 1
Neutrophil count decreased (Investigations) | 0 | 0 | 1
White blood cell count decreased (Investigations) | 0 | 0 | 1
Back pain (Musculoskeletal and connective tissue disorders) | 5 | 2 | 2
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 | 0 | 1
Muscle spasms (Musculoskeletal and connective tissue disorders) | 0 | 1 | 1
Muscle weakness (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0
Neck pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1
Hypoesthesia (Nervous system disorders) | 3 | 2 | 0
Sciatica (Nervous system disorders) | 2 | 0 | 1
Headache (Nervous system disorders) | 2 | 0 | 0
Areflexia (Nervous system disorders) | 0 | 0 | 1
Hyporeflexia (Nervous system disorders) | 0 | 0 | 1
Migraine (Nervous system disorders) | 0 | 0 | 1
Radiculopathy (Nervous system disorders) | 1 | 0 | 0
Sensory loss (Nervous system disorders) | 0 | 0 | 1
Upper respiratory tract infection (Infections and infestations) | 1 | 1 | 1
Urinary tract infection (Infections and infestations) | 0 | 1 | 2
COVID-19 (Infections and infestations) | 2 | 0 | 0
Rhinitis (Infections and infestations) | 1 | 0 | 0
Pain (General disorders) | 5 | 0 | 1
Injection site pain (General disorders) | 2 | 1 | 0
Gait disturbance (General disorders) | 0 | 0 | 1
Malaise (General disorders) | 0 | 0 | 1
Anemia (Blood and lymphatic system disorders) | 0 | 1 | 1
Leukopenia (Blood and lymphatic system disorders) | 1 | 0 | 1
Neutropenia (Blood and lymphatic system disorders) | 1 | 0 | 1
Increased tendency to bruise (Blood and lymphatic system disorders) | 1 | 0 | 0
Limb injury (Injury, poisoning and procedural complications) | 1 | 1 | 0
Back injury (Injury, poisoning and procedural complications) | 0 | 0 | 1
Rib fracture (Injury, poisoning and procedural complications) | 0 | 0 | 1
Vaccination complication (Injury, poisoning and procedural complications) | 1 | 0 | 0
Abdominal adhesions (Gastrointestinal disorders) | 1 | 0 | 0
Diarrhea (Gastrointestinal disorders) | 1 | 0 | 0
Nausea (Gastrointestinal disorders) | 0 | 0 | 1
Small intestinal obstruction (Gastrointestinal disorders) | 1 | 0 | 0
Anxiety (Psychiatric disorders) | 0 | 2 | 0
Abnormal dreams (Psychiatric disorders) | 1 | 0 | 0
Depression (Psychiatric disorders) | 0 | 0 | 1
Hypernatremia (Metabolism and nutrition disorders) | 0 | 0 | 1
Iron deficiency (Metabolism and nutrition disorders) | 0 | 0 | 1
Dermatitis contact (Skin and subcutaneous tissue disorders) | 0 | 0 | 1
Erythema (Skin and subcutaneous tissue disorders) | 0 | 0 | 1
Pruritis (Skin and subcutaneous tissue disorders) | 1 | 0 | 0
Proteinuria (Renal and urinary disorders) | 0 | 0 | 1
Renal colic (Renal and urinary disorders) | 0 | 0 | 1
Menopausal symptoms (Reproductive system and breast disorders) | 0 | 0 | 1

LIMITATIONS AND CAVEATS:
Due to the impact of COVID-19 and associated enrollment difficulties, the study was terminated with a total sample size of 56 randomized patients.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2020-06-17): https://cdn.clinicaltrials.gov/large-docs/77/NCT03952377/Prot_002.pdf
  • Statistical Analysis Plan (2022-07-13): https://cdn.clinicaltrials.gov/large-docs/77/NCT03952377/SAP_003.pdf